CLINICAL TRIAL: NCT06727851
Title: Quality Improvement in Endoscopy: Has the Implementation of the ESGE Guideline 2017 Led to a Reduction in Post-ERCP Pancreatitis? A Multicenter Trial
Brief Title: ESGE-Quality Improvement in Endoscopy: ERCP
Acronym: QIC_ERCP
Status: Enrolling by invitation | Type: Observational
Sponsor: Universität Münster (Other)
Collaborators: University of Kiel (Other); University of Copenhagen (Other); Johannes Gutenberg University Mainz (Other); University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: Quality improvement in ERCP
Record Dates: First submitted 2024-11-28; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: performance measures; ESGE; post-ERCP pancreatitis; quality in endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group before introduction of the QIC-initiative (before 2017): The study shall provide the investigators with information whether the introduction of the quality performance measures adopted by the European Society of Gastrointestinal Endoscopy (ESGE) will actually lead to an improvement in quality. The study will compare the quality development in endoscopy based on following time intervals: 1. before introduction of the QIC-initiative (before 2017) 2. after the introduction of the initiative (2017-2023) (both retrospective data) 3. prospectively, from 2024 onwards. The focus of this study we will be the key performance indicator post-ERCP pancreatitis (PEP). In the ESGE-guideline, a minimum standard of <10% and a target standard of <5% was recommended. Different studies described the incidence of post-ERCP pancreatitis between 3,47% and 10,2%.
- Group after introduction of the QIC-initiative (2017-2023): The study shall provide the investigators with information whether the introduction of the quality performance measures adopted by the European Society of Gastrointestinal Endoscopy (ESGE) will actually lead to an improvement in quality. The study will compare the quality development in endoscopy based on following time intervals: 1. before introduction of the QIC-initiative (before 2017) 2. after the introduction of the initiative (2017-2023) (both retrospective data) 3. prospectively, from 2024 onwards. The focus of this study we will be the key performance indicator post-ERCP pancreatitis (PEP). In the ESGE-guideline, a minimum standard of <10% and a target standard of <5% was recommended. Different studies described the incidence of post-ERCP pancreatitis between 3,47% and 10,2%.
- Prospective Group: The study shall provide the investigators with information whether the introduction of the quality performance measures adopted by the European Society of Gastrointestinal Endoscopy (ESGE) will actually lead to an improvement in quality. The study will compare the quality development in endoscopy based on following time intervals: 1. before introduction of the QIC-initiative (before 2017) 2. after the introduction of the initiative (2017-2023) (both retrospective data) 3. prospectively, from 2024 onwards. The focus of this study we will be the key performance indicator post-ERCP pancreatitis (PEP). In the ESGE-guideline, a minimum standard of <10% and a target standard of <5% was recommended. Different studies described the incidence of post-ERCP pancreatitis between 3,47% and 10,2%.

SUMMARY:
The primary aim of the present study is to compare the incidence of post-ERCP pancreatitis (PEP) before and after the implementation of the QIC-guideline in 2017: "Performance measures for ERCP and endoscopic ultrasound: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative".

DETAILED DESCRIPTION:
In 2017, a new guideline addressing the quality in ERCP entitled "Performance measures for ERCP and endoscopic ultrasound: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative" was published. The focus of the quality improvement committee (QIC) of the ESGE is to ensure high standard of all endoscopy examinations throughout Europe by adhering to quality-improving factors (key performance indicators and minor performance indicators as defined by the ESGE).

The study shall provide the investigators with information whether the introduction of the quality performance measures adopted by the European Society of Endoscopy (ESGE) will actually lead to an improvement in quality.

The study will compare the quality development in endoscopy based on following time intervals:

1. before introduction of the QIC-initiative (before 2017)
2. after the introduction of the initiative (2017-2023) (both retrospective data),
3. prospectively, from 2024 onwards.

The primary endpoint of this study will be the key performance indicator post-ERCP pancreatitis (PEP). In the ESGE-guideline, a minimum standard of <10% and a target standard of <5% was recommended. Different studies described the incidence of post-ERCP pancreatitis between 3,47% and 10,2%.

The investigators hope that this study will lead to even greater patient safety in the future by improving findings and examination quality and therefore reduce the incidence of post-ERCP pancreatitis. In addition, the aim is to harmonize the high endoscopic standards throughout Europe.

ELIGIBILITY:
Inclusion Criteria:nclusion criteria Individuals eligible for inclusion are patients referred for ERCP who do not fulfill one of the following exclusion criteria

Exclusion criteria

* Individuals eligible for inclusion are patients referred for ERCP who do not fulfill one of the following exclusion criteria
* Age under 18 years
* Inability to understand information for participation
* Refusal of participation, missing cooperativity, e.g., due to age or disease
* Pregnant or lactating patients
* Patients with > 1 ERCP during the hospital stay: only the initial ERCP will be evaluated

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals eligible for inclusion are patients referred for ERCP who do not fulfill one of the following exclusion criteria
  * Age under 18 years
  * Inability to understand information for participation
  * Refusal of participation, missing cooperativity, e.g., due to age or disease
  * Pregnant or lactating patients
  * Patients with > 1 ERCP during the hospital stay: only the initial ERCP will be evaluated
Sampling Method: Non-Probability Sample
Enrollment: 1254 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis (PEP) | 2016 - 2025
  Comparison of the incidence of PEP before and after the implementation of the guideline. i. Clinical illness with typical pain (physical examination: pain in the upper belly with/without radiation to the back, tenderness when touching the belly) ii. laboratory testing with 3x increase of lipase (or amylase) iii. Characteristic findings in CE-CT, MRI or transabdominal sonography iv. Requiring extension of hospital stay

SECONDARY OUTCOMES:
Adequate antibiotic prophylaxis before ERCP | 2016 - 2025
  Rate of adequate antibiotic prophylaxis before ERCP
Bile duct cannulation | 2016 - 2025
  Rate of successful bile duct cannulation
Appropriate stent placement in patients with biliary obstruction below the hilum | 2016 - 2025
  Rate of appropriate stent placement in patients with biliary obstruction below the hilum
Bile duct stone extraction | 2016 - 2025
  Rate of successful bile duct stone extraction

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Domagk, MD, Principal Investigator — Universität Münster
Locations (1):
- University of Muenster, Josephs Hospital Warendorf, Academic Teaching Hospital, Warendorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akshintala VS, Kanthasamy K, Bhullar FA, Sperna Weiland CJ, Kamal A, Kochar B, Gurakar M, Ngamruengphong S, Kumbhari V, Brewer-Gutierrez OI, Kalloo AN, Khashab MA, van Geenen EM, Singh VK. Incidence, severity, and mortality of post-ERCP pancreatitis: an updated systematic review and meta-analysis of 145 randomized controlled trials. Gastrointest Endosc. 2023 Jul;98(1):1-6.e12. doi: 10.1016/j.gie.2023.03.023. Epub 2023 Mar 31. PMID 37004815
- [Background] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Domagk D, Oppong KW, Aabakken L, Czako L, Gyokeres T, Manes G, Meier P, Poley JW, Ponchon T, Tringali A, Bellisario C, Minozzi S, Senore C, Bennett C, Bretthauer M, Hassan C, Kaminski MF, Dinis-Ribeiro M, Rees CJ, Spada C, Valori R, Bisschops R, Rutter MD. Performance measures for ERCP and endoscopic ultrasound: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2018 Nov;50(11):1116-1127. doi: 10.1055/a-0749-8767. Epub 2018 Oct 19. PMID 30340220